CLINICAL TRIAL: NCT07335861
Title: Evaluation of the Efficacy of Hyalomatrix® in the Healing of Chronic Venous Leg Ulcers: A Randomized Controlled Multicenter Crossover Trial
Brief Title: Evaluation of the Efficacy of Hyalomatrix® in the Healing of Chronic Venous Leg Ulcers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NuScience Medical Biologics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HALO
Record Dates: First submitted 2026-01-09; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Venous Leg Ulcer; Chronic Wounds
MeSH Terms: conditions — Varicose Ulcer | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The subject will be randomized to one of the following treatments:
  Standard of care (SOC) combined with Hyalomatrix or SOC alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care (Active Comparator): Wound cleansing, sharps debridement, dressing for moisture balance, and compression therapy
  Interventions: Other: Standard of Care
- Hyalomatrix + Standard of Care (Experimental): Wound cleansing, sharps debridement, Hyalomatrix application, dressing for moisture balance, compression therapy
  Interventions: Device: Hyalomatrix

INTERVENTIONS:
Device: Hyalomatrix — Hyalomatrix is a hyaluronic acid-based wound dressing designed for advanced wound therapy.
  Arms: Hyalomatrix + Standard of Care
Other: Standard of Care — Wound cleansing, Sharps debridement, Dressing for moisture balance, Compression therapy
  Other Names: SOC
  Arms: Standard of Care

SUMMARY:
This is a randomized controlled trial evaluating the efficacy of HYALOMATRIX in conjunction with standard of care vs. standard of care alone in treating venous leg ulcers.

DETAILED DESCRIPTION:
This research will take place across multiple medical centers, where both researchers and participants will know which treatment is being used (open label). Patients who agree to participate and meet the study requirements during screening will be randomly assigned to one of two groups: either standard of care (SOC) alone, or SOC plus Hyalomatrix. The study includes a crossover component for subjects in the SOC arm. At treatment visit 13 (approximately 84 days post-randomization), SOC arm subjects not having achieved complete wound closure, and still meeting the inclusion/exclusion criteria, are eligible to crossover to the IP arm (SOC plus Hyalomatrix). Crossover subjects will begin IP arm treatment with weekly Hyalomatrix applications for up to 12 treatment visits. The subject will continue follow-up per the original schedule. As this is a post-marketing study, it will gather information regarding the efficacy of treatment while also supporting insurance reimbursement decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 18 years of age or older
2. Subject has a medical diagnosis of venous leg ulcer or venous insufficiency with a lower extremity wound
3. Subject has a venous leg ulcer present for 4 weeks or greater (documented in medical record), and less than 12 months duration if being treated with continuous SOC
4. Subject has a venous leg ulcer with a historical wound measurement showing less than 25% healing within 14 days prior to screening
5. Subject has a venous leg ulcer with screening wound measurement showing less than 25% healing within 14 days prior to randomization
6. Subject has a venous leg ulcer without infection or clinically visible exposed bone
7. Index wound is a minimum of 1 cm2 and a maximum of 30 cm2 at first treatment visit
8. Adequate circulation if wound is location on the lower extremity demonstrated by an ABI of >0.7 and <1.3, or TBI of >0.6 within 30 days prior to informed consent OR an arterial ultrasound noted with patent circulation and without significant stenosis 90 days prior to the first treatment visit.
9. Venous Leg Ulcer is being treated with compression therapy for 14 days prior to treatment visit 1
10. Index wound is free of necrotic debris prior to Hyalomatrix application
11. Female subjects of childbearing potential having a negative pregnancy test prior to randomization
12. Index wound is free of infection prior to randomization and during screening phase noted with the NERDS Assessment. Infection must be adequately treated and controlled prior to randomization.
13. Subject is able and willing to follow the protocol requirements
14. Subject had signed informed consent
15. If 2 or more wounds are present, the wounds must be separated by at least 2 cm

Exclusion Criteria:

1. Subject does not have a diagnosis of venous leg ulcer or venous insufficiency with a wound located on the lower extremity
2. Subject has a known life expectancy of <1 year
3. Subject is unable to comply with protocol treatment
4. Subject has comorbid conditions that may compromise subject safety or wound healing in the opinion of the investigator, such as serious cardiovascular, renal, liver, pulmonary, autoimmune, palliative care, or inherited blood disorders
5. Subject actively being treated for malignant disease or history of malignancy or radiation therapy at the site of wound
6. Subject has comorbid conditions that may compromise subject safety in the opinion of the investigator
7. Known contraindications to tissue-engineered allograft
8. Concurrent participation in alternative clinical trial that involves investigational drug or HCT/P interfering with wound treatment and/or healing.
9. Subject is pregnant or breastfeeding
10. Subject with history of immunosuppressant treatment (systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or topical steroid application to the wound surface for >2 weeks duration within 30 days prior to randomization; or anticipated use of the above during the course of the study
11. Wound previously treated with CAMPs, tissue engineered, or scaffold materials within 30 days prior to randomization
12. Venous leg ulcer with active infection
13. Wound depth with visible exposed bone
14. HBOT within 14 days prior to randomization
15. Revascularization surgery on the index wound leg within 30 days of screening phase
16. Index wound suspicious of neoplasm in the opinion of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Wound Closure | 1-12 weeks
  The primary endpoint will be the percentage of target wounds that achieve complete wound closure within 12 weeks.

SECONDARY OUTCOMES:
Weekly Percentage Area Reduction | 1-12 weeks
  The percentage reduction in wound area from 1-12 weeks will be measured weekly using digital photographic planimetry and physical examination.
Pain Assessment | 1-14 weeks
  Change in pain associated with the target wound will be assessed using the Numeric Pain Rating Scale throughout the study. Numeric Rating on a scale of 0-10. o is No pain and 10 is the worst possible pain.

OTHER OUTCOMES:
Time to Closure | 1-12 weeks
  Average number of grafts/weeks used to achieve wound closure
Follow-Up Closure | 2 weeks
  Number of wounds that re-opened during the 2-week follow-up
Adverse Events and Serious Adverse Events | 1-12 weeks
  The number and nature of adverse events (AEs) and serious adverse events (SAEs) occurring during the study will be tracked and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Angelina Ferguson, DNP, Study Director — SygNola, LLC

IPD SHARING:
Plan to Share IPD: No